CLINICAL TRIAL: NCT06309589
Title: Department of Infectious Diseases, People's Hospital of Xinjiang Uygur Autonomous Region
Brief Title: The Effectiveness of Combining Ursodeoxycholic Acid With Vitamin D in Treating Patients With Primary Biliary Cholangitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yilihamu·Abilitifu (Other)
Responsible Party: Sponsor-Investigator, Yilihamu·Abilitifu, People's Hospital of Xinjiang Uygur Autonomous Region, People's Hospital of Xinjiang Uygur Autonomous Region
Organization: People's Hospital of Xinjiang Uygur Autonomous Region (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YIHM
Record Dates: First submitted 2024-03-01; First posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Primary Biliary Cholangitis
Keywords: Primary biliary cholangitis; Ursodeoxycholic acid; Vitamin D
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — Vitamin D; Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): experimental group received UDCA(Losan Pharma GmbH, registration number H20181059, 13-15 mg/day/kg) combined with Vitamin D3 (1200 IU per day) treatment for 1year
  Interventions: Drug: Vitamin D
- control group (No Intervention): control group received UDCA(Losan Pharma GmbH, registration number H20181059, 13-15 mg/day/kg) treatment for 1 year

INTERVENTIONS:
Drug: Vitamin D — experimental group received UDCA combined with vitamin D3 (1200 IU per day) treatment
  Other Names: Vitamin D3
  Arms: experimental group

SUMMARY:
The goal of this clinical trial is to compare in the effectiveness of combining ursodeoxycholic acid and vitamin D in treating patients with primary biliary cholangitis.

DETAILED DESCRIPTION:
A prospective analysis will be conducted on 60 patients with primary PBC who were admitted to our Infectious Diseases Department and outpatient clinic. All patients will take UDCA capsules orally and divide into two groups: the experimental group, which received UDCA combined with Vitamin D(1200 IU per day) treatment, and the control group. The control group will receive UDCA treatment alone for one year, selected through a random number table method. After one year, the control group will be further divided into two groups using the same method. One group will continue to receive UDCA alone, while the other will receive a combination of UDCA and vitamin D for an additional year. Clinical data, clinical manifestations, blood tests, and imaging tests will be collected during the initial and subsequent treatments. The efficacy will be evaluated using the Paris I and Barcelona standards.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must meet the diagnostic criteria for PBC ;
2. The patient must have been diagnosed at the age of 18 or older;
3. The patient must have completed at least 2 years of treatment and have complete and accessible clinical data;
4. The patient must have strictly followed the doctor's prescription during the treatment period and not have interrupted the treatment arbitrarily.

Exclusion Criteria:

1. The study excluded patients with autoimmune hepatitis or primary sclerosing cholangitis.
2. Patients with other acute and chronic liver diseases were also excluded.
3. Patients with serious cardiopulmonary diseases were excluded as well.
4. Pregnant or lactating women were not included in the study.
5. Patients who randomly interrupted or adjusted their medication during the treatment period were excluded.
6. Patients who lacked follow-up were also excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
UDCA response: Paris I criteria | 1 year
  The ALP levels should be no more than three times the upper limit of normal (3xULN), while the AST levels should be no more than two times the ULN, and bilirubin levels should be normal after one year of standard treatment.
UDCA response: Barcelona criteria | 1 year
  After one year of standard treatment, the ALP levels should decrease by more than 40% or reach normal levels.

CONTACTS AND LOCATIONS:
Overall Officials: Nanfang Li, Prof., Principal Investigator — People's Hospital of Xinjiang Uygur Autonomous Region
Locations (1):
- People's Hospital of Xinjiang Uygur Autonomous Region, Ürümqi, Xinjiang, China

IPD SHARING:
Plan to Share IPD: No